CLINICAL TRIAL: NCT06023550
Title: Analysis of Complicated Infections in Pediatric and Adult Populations Treated by Otorhinolaryngologist
Brief Title: Complicated Infections in Otorhinolaryngology
Acronym: ENT_infect
Status: Recruiting | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Domen Vozel, MD, PhD, Domen Vozel, MD, PhD, ENT specialist, University Medical Centre Ljubljana
Other Study IDs: ENT infections
Record Dates: First submitted 2023-08-27; First posted 2023-09-05 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Sinusitis; Otitis; Laryngitis; Lymphadenitis; Quinsy; Peritonsillar Abscess; Parapharyngeal Abscess; Preseptal Cellulitis; Subperiosteal Abscess; Orbital Abscess; Epiglottitis
MeSH Terms: conditions — Sinusitis; Otitis; Laryngitis; Lymphadenitis; Peritonsillar Abscess; Orbital Cellulitis; Epiglottitis | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Complicated sinonasal infection: Group of patients with a complicated sinonasal infection, including local or systemic complications.
  Interventions: Other: Treatment with surgery and/or conservative measures
- Complicated ear or temporal bone infection: Group of patients with a complicated ear or temporal bone infection, including local or systemic complications.
  Interventions: Other: Treatment with surgery and/or conservative measures
- Complicated neck soft tissue infection: Group of patients with a complicated neck soft tissue infection, including local or systemic complications.
  Interventions: Other: Treatment with surgery and/or conservative measures
- Complicated laryngeal infection: Group of patients with a complicated laryngeal infection, including local or systemic complications.
  Interventions: Other: Treatment with surgery and/or conservative measures

INTERVENTIONS:
Other: Treatment with surgery and/or conservative measures — Patients will be treated according to established clinical practice with surgery and/or conservative measures.

SUMMARY:
This observational study aims to learn more about complicated infections treated by otorhinolaryngologists. The main questions to answer are:

* What is the management of complicated sinonasal infections in Ljubljana, Slovenia,
* What is the management of complicated ear and temporal bone infections in Ljubljana, Slovenia,
* What is the management of complicated neck soft tissue infections in Ljubljana, Slovenia,
* What is the management of complicated laryngeal infections in Ljubljana, Slovenia

Participants will receive standard treatment according to the established evidence-based clinical practice.

DETAILED DESCRIPTION:
The main purpose of the research is to obtain own data on the treatment of patients with infections in ENT areas that require targeted treatment by an otolaryngologist at the hospital level. Based on these results, treatment outcome would be improved and hospitalization time would be shortened. We would establish clinical pathways for the treatment of these diseases in Slovenia. There is still no data on the treatment of these diseases in ENT departments in Slovenia, so one of the main purposes of the research is to obtain objective indicators of the success of treatment in comparison with other countries and a rough epidemiological assessment of the disease in Slovenia.

The research would establish a database of patients with complicated infections in ENT areas at the University Clinical Center Ljubljana, which would be used for prospective analysis even after the research was completed. The register would also enable transparency in the treatment of these patients in the future.

The main questions to answer are:

* What is the management of complicated sinonasal infections in Ljubljana, Slovenia,
* What is the management of complicated ear and temporal bone infections in Ljubljana, Slovenia,
* What is the management of complicated neck soft tissue infections in Ljubljana, Slovenia,
* What is the management of complicated laryngeal infections in Ljubljana, Slovenia

Participants will receive standard treatment according to the established evidence-based clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses: rhinitis AND/OR sinusitis AND/OR facial cellulitis AND/OR facial abscess AND/OR nasal furuncle AND/OR infection of the outer AND/OR middle AND/OR inner ear AND/OR temporal bone AND/OR infection of the soft tissues of the neck with/without bone and cartilage involvement AND/OR laryngitis AND/OR epiglottitis (or supraglottitis) AND/OR
* complication of inflammation of the nose and paranasal cavities AND/OR ear AND/OR temporal bone AND/OR:
* treated at the Department of Otorhinolaryngology and Cervicofacial Surgery, University Medical Center Ljubljana.

Exclusion Criteria:

* disagreement of the patient and/or parents (or legal guardians) with inclusion in the research,
* failure to meet the inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with complicated infections treated by otorhinolaryngologists in the tertiary otorhinolaryngology referral centre.
Sampling Method: Non-Probability Sample
Enrollment: 2550 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 12 months
  Number of living patients without a disease

CONTACTS AND LOCATIONS:
Overall Officials: Domen Vozel, MD, PhD, Principal Investigator — Department of Otorhinolaryngology and Cervicofacial Surgery, UMC Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No